CLINICAL TRIAL: NCT06416163
Title: A Prospective Observational Study Investigating Whether Nocturnal Hypoxaemia and Exercise Induced Desaturation Predict Functional Deterioration in Patients With Fibrotic Interstitial Lung Disease
Brief Title: FIBRotic Interstitial Lung Disease With Nocturnal hypOXaemia and EXercise Induced desaTuRAtion
Acronym: FIBRINOX-EXTRA
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 329843
Record Dates: First submitted 2024-01-19; First posted 2024-05-16 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Interstitial Lung Disease; Fibrosis Lung; Pulmonary Hypertension
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Hypertension, Pulmonary | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective: All participants will be in one group which is the collection of retrospective data
  Interventions: Other: Prospective

INTERVENTIONS:
Other: Prospective — Collection of prospective data all ready available for participant

SUMMARY:
This is an observational clinical research study investigating patients with fibrotic interstitial lung disease (fILD), also known as pulmonary fibrosis.

It is not known why some patients with fILD clinically deteriorate. This study will investigate whether measuring oxygen levels during sleep or exercise can help identify patients who are at increased risk of clinical deterioration.

DETAILED DESCRIPTION:
This work will build upon the FIBRINOX study, previous clinical research conducted by the Guy's and St Thomas' ILD research team. The FIBRINOX study showed that patients with fILD and normal oxygen saturations at rest, but who desaturate whilst asleep or during exercise, have a significantly increased mortality and greater reduction in quality of life compared to patients who do not desaturate at night or during exercise.

The reasons for these differences in mortality and health related quality of life are not known. Data suggests that worsening fILD and the development of pulmonary hypertension, a condition characterised by increased pressure in the pulmonary arteries that is associated with poorer outcomes, may be playing a role.

This clinical research study will recruit approximately 160 patients with a tertiary ILD centre diagnosis of fibrotic interstitial lung disease (fILD). Data from routinely performed investigations as part of tertiary ILD assessment will be systematically recorded.

Investigations will include lung function tests, echocardiography, blood tests, a 6-minute walk test and overnight oximetry. Participants will also complete several quality-of-life questionnaires. These investigations will be performed at baseline, and again at 12 months, with all tests also repeated at 6 months except for an echocardiogram. After the initial 1 year study period, a 3 year post-recruitment mortality and right heart catheter check will be performed using the participants' medical records. Data will be collected from CT scans and right heart catheters if performed during the study period as part of the participants usual clinical care.

This study is designed to establish whether patients with fILD who desaturate during sleep or exercise are more likely to experience functional decline, as well as confirm previous findings of increased mortality and worsening quality of life as demonstrated in the FIBRINOX study. The data generated by this observational study will help generate future hypotheses, research questions and clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 year and over
2. Tertiary MDT diagnosis of FILD with >10% fibrosis on CT chest as determined by the investigator. Underlying diagnoses to include but not limited to: idiopathic pulmonary fibrosis (IPF), non-specific interstitial pneumonitis (NSIP), chronic hypersensitivity pneumonitis (CHP), connective tissue disease-related interstitial lung disease (CTD-ILD), fibrotic organising pneumonia (FOP) and pulmonary sarcoidosis.
3. Able to provide informed written consent

Exclusion Criteria:

1. The use of or any indication for long-term oxygen therapy (LTOT)
2. Known moderate or severe obstructive sleep apnoea with an apnoea/hypopnoea index (AHI) or oxygen desaturation index (ODI) over 15 events per hour
3. Radiological predominance of emphysema compared with fibrosis on CT chest
4. Inability to complete all health status questionnaires as set out in this protocol, with appropriate support
5. A confirmed diagnosis of pulmonary hypertension
6. Significant cardiovascular comorbidity including severe, uncontrolled hypertension, uncontrolled arrhythmia, recent acute coronary syndrome within 30 days prior to study enrolment, that could mean exercise testing poses a risk to patient health, in the opinion of the investigator
7. Musculoskeletal comorbidity that will preclude the participant's ability to reliably complete the complete 6-minute walk test (6MWT)
8. Participation in another research project which may confound this study's research findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a tertiary ILD centre diagnosis of fibrotic interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | 52 weeks
  As measured by 6-minute walk test

SECONDARY OUTCOMES:
Mortality | 52 and 156 weeks
  If death occurs during the study period, and the cause of death
Clinical deterioration | 52 weeks
  Defined by: decline in forced vital capacity (FVC) >10% or death
Decline in FVC | 52 weeks
  Decline in forced vital capacity
Decline in TLCO | 52 weeks
  Decline in total diffusing capacity of the lungs for carbon monoxide
Pulmonary hypertension | 52 and 156 weeks
  Right heart catheter confirmed pulmonary hypertension
Change in arterialised capillary blood gas pO2 | 52 weeks
  Arterialised capillary blood gas partial pressure of oxygen
Change in arterialised capillary blood gas oxygen saturations | 52 weeks
  Arterialised capillary blood gas oxygen saturations
Change in arterialised capillary blood gas pCO2 | 52 weeks
  Arterialised capillary blood gas partial pressure of carbon dioxide
Change in arterialised capillary blood gas HCO3 | 52 weeks
  Arterialised capillary blood gas partial pressure of bicarbonate
Change in arterialised capillary blood gas pH | 52 weeks
  Arterialised capillary blood gas pH
Time to first acute exacerbation of fILD | 52 weeks
  The number of days until the participant requires hospital admission for an acute worsening of their respiratory condition, not attributable to other causes
Rate of acute exacerbation of fILD | 52 weeks
  The number of times the participant requires hospital admission for an acute worsening of their respiratory condition, not attributable to other causes
Change in NT-proBNP/BNP level | 52 weeks
  Change in NT-proBNP/BNP level from baseline
Change in troponin level | 52 weeks
  Change in troponin level from baseline
Change in peak TRV | 52 weeks
  Change in peak tricuspid regurgitation velocity (TRV)
Change in cardiac chamber size/area | 52 weeks
  Change in cardiac chamber size/area
Change in cardiac chamber area | 52 weeks
  Change in cardiac chamber area
Change in RV/LV basal diameter area ratio | 52 weeks
  Change in right ventricle to left ventricle basal diameter area ratio
Change in MPA:AA diameter ratio | 52 weeks
  Change in main pulmonary artery to ascending aorta diameter ratio
Change in TAPSE/sPAP ratio | 52 weeks
  Change in tricuspid annular plane systolic excursion to systolic pulmonary artery pressure ratio
Change in European Quality of Life 5-Dimensions 5-Levels (EQ-5D-5L) questionnaire score | 52 weeks
  Change in score of European Quality of Life 5-Dimensions 5-Levels (EQ-5D-5L) questionnaire
Change in King's Brief Interstitial Lung Disease (KBILD) questionnaire score | 52 weeks
  Change in score of King's Brief Interstitial Lung Disease (KBILD) questionnaire
Change in Living with Pulmonary Fibrosis (L-IPF) questionnaire score | 52 weeks
  Change in score of Living with Pulmonary Fibrosis (L-IPF) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alex West, MBBS, Principal Investigator — Guys and St. Thomas NHS Foundation Hospital
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared or made available to researchers outside of the site research team where the patient is based, and GSTT ILD research team.

REFERENCES:
- [Background] Myall KJ, West AG, Martinovic JL, Lam JL, Roque D, Wu Z, Maher TM, Molyneaux PL, Suh ES, Kent BD. Nocturnal Hypoxemia Associates With Symptom Progression and Mortality in Patients With Progressive Fibrotic Interstitial Lung Disease. Chest. 2023 Nov;164(5):1232-1242. doi: 10.1016/j.chest.2023.05.013. Epub 2023 May 13. PMID 37187434